CLINICAL TRIAL: NCT06507332
Title: Combination Letrozole and Clomiphene Citrate Versus Letrozole Alone for Ovulation Induction in Women With Polycystic Ovary Syndrome: A Randomized Control Trial
Brief Title: Combination Letrozole and Clomiphene Citrate Versus Letrozole Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed Adel Mousa
Record Dates: First submitted 2024-07-07; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Letrozole group) (Active Comparator): About 32 patients will receive letrozole 2.5 mg tablets only , once daily from the third date of the menses for 5 days for 3 successive periods
  Interventions: Drug: Letrozole 2.5mg
- Group 2 (Letrozole and Clomiphene Citrate) (Active Comparator): About 32 patients will receive combined letrozole 2.5 mg tablets once daily and clomiphene citrate 50 mg tablets once daily from the third date of the menses for 5 days for 3 successive periods
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Letrozole 2.5mg — to assess and compare the efficacy of Combination of letrozole and clomiphene citrate versus letrozole alone for ovulation induction in women with polycystic ovary syndrome (PCOS)
  Other Names: Clomiphene Citrate

SUMMARY:
Clomiphene citrate is a non-steroidal triphenylethylene derivative distantly related to diethylstilbestrol. It acts as a selective estrogen receptor modulator (SERM), similar to tamoxifen and raloxifene. All three drugs are competitive inhibitors of estrogen binding to estrogen receptors (ERs) and have mixed agonist and antagonist activity, depending upon the target tissue.

Letrozole is a potent, nonsteroidal, aromatase inhibitor, originally used for postmenopausal breast cancer therapy.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in reproductive-age women and the most common cause of anovulatory infertility. The treatment of infertility in patients with PCOS focuses on ovulation induction. Many treatment regimens have been used, with varying success, to achieve ovulation, pregnancy, and live birth.

Clomiphene citrate (CC) is a commonly prescribed pharmacologic agent used to induce ovulation in women with PCOS. It works as a selective estrogen receptor modulator by competitively attaching to nuclear estrogen receptors. As the negative feedback of estrogen is reduced, secretion of gonadotropin hormones increases, inducing ovarian follicular growth.

Clomiphene citrate (CC) also has an anti-estrogenic effect on endometrial development and cervical mucus production,which has been suggested to contribute to a relatively low pregnancy rate despite a high ovulation rate.

Letrozole is another commonly used oral ovulation induction agent, with a different mechanism of action. It works as a highly selective aromatase inhibitor, preventing androgen-to-estrogen conversion. One proposed mechanism is via suppressed estrogen production resulting in decreased negative feedback on the hypothalamus and increased secretion of Follicular Stimulating Hormone (FSH). An additional proposed mechanism of improved ovulatory rates with the use of letrozole is increased follicular sensitivity to FSH resulting from temporarily increased intraovarian androgens .

Letrozole may offer a benefit over CC for ovulation induction because it does not block estrogen receptors in both central and peripheral target tissues, and normal central feedback mechanisms remain intact. The Pregnancy and Polycystic Ovary Syndrome (PPCOS) trial, a randomized controlled trial comparing letrozole and CC, demonstrated that letrozole was associated with a higher live birth rate (27.5% vs. 19.1%; P=007; rate ratio 1.44, 95% confidence interval [CI] 1.10-1.87) and cumulative ovulation rate (61.7% vs. 48.3%; P<.001) among women with PCOS.

Other than letrozole or CC for ovulation induction, there are few treatment options available to PCOS patients except proceeding to gonadotropin injections or in vitro fertilization, both of which are associated with increased cost and risk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infertility, defined as the inability of couple to achieve a pregnancy after 12 months of regular timed unprotected intercourse in women <35 years of age or after 6 months in women >35 years of age.
* Diagnosis of PCOS based on the Rotterdam criteria, including two of the following three findings: oligomenorrhea or chronic anovulation, hyperandrogenism (clinical or laboratory), and polycystic ovary(ies) on ultrasound .
* Normal HSG
* Normal semen analysis.
* Has capacity to participate in the study.

Exclusion Criteria:

* Unexplained infertility.
* Other conditions that can cause chronic anovulation and androgen excess such as hyperthyroidism by thyroid profile.
* congenital adrenal hyperplasia
* Cushing
* Untreated hyperprolactinemia.
* Medical conditions not well controlled or contraindicated to get pregnant with it like (uncontrolled diabetes mellitus, hypertension) .
* endometrial hyperplasia/cancer
* Allergy or contraindications to letrozole or CC. (by history)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Check | 2 weeks after ovulation
  The participants required to make pregnancy test after Receiving the drugs of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dina Yahia, Professor, Study Chair — Department of Obstetrics & Gynecology,Ain Shams University; Al Hassan Mohammad Khedr, Lecturer, Study Director — Department of Obstetrics & Gynecology,Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided